CLINICAL TRIAL: NCT04043039
Title: Platelet Rich Fibrin in the Treatment of Palatal Wounds After Full Thickness Palatal Grafts Harvesting: A Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin in the Treatment of Full Thickness Palatal Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Head of Periodontology, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 072019
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FULL THICKNESS PALATAL GRAFT (Experimental): the full thickness palatal wound will be protected by a quadruple layer of Platelet Rich Fibrin obtained by folding on itself 2 Platelet Rich Fibrin membrane or by gelatine sponge
  Interventions: Procedure: Palatal wound bandage with PRF; Procedure: Palatal wound bandage with Gelatine Sponge
- FREE GINGIVAL GRAFT (Active Comparator): the Epithelialized Free Gingival Grafts palatal wound will be protected by a quadruple layer of Platelet Rich Fibrin obtained by folding on itself 2 Platelet Rich Fibrin membrane or by gelatine sponge
  Interventions: Procedure: Palatal wound bandage with PRF; Procedure: Palatal wound bandage with Gelatine Sponge

INTERVENTIONS:
Procedure: Palatal wound bandage with PRF — palatal wound will be protected by a quadruple layer of Platelet Rich Fibrin obtained by folding on itself 2 Platelet Rich Fibrin membranes
Procedure: Palatal wound bandage with Gelatine Sponge — palatal wound will be protected by gelatine sponge

SUMMARY:
In this study it will be investigated the usefulness of Platelet-Rich Fibrin (PRF) on in the full thickness palatal graft donor site healing acceleration and in the patient's morbidity reduction. Eighty patients, with at least one gingival recession will be treated by a flap with connective tissue graft(CTG). In the test group (20 patients) and in the control group 2 a quadruple layer of PRF membrane will be placed over the palatal wounds; conversely, the control groups 2-4 patients will be treated by an absorbable gelatin sponge. Patients will be monitored at 1, 2, 3 and 4 weeks after surgery for the complete re-epithelialization of the palatal wound (CWE), the alteration of sensibility (AS) around the wound area, the post-operative discomfort (D), and the changes of feeding habits (CFH) by a visual analogic scale (VAS) evaluation. Furthermore, the analgesics consumption and the existence of delayed bleeding from the palatal wound (DWB) during the first post-operative week will be assessed.

DETAILED DESCRIPTION:
In this study it will be investigated the usefulness of Platelet-Rich Fibrin (PRF) on in the full thickness palatal graft donor site healing acceleration and in the patient's morbidity reduction. Eighty patients, with at least one gingival recession will be treated by a coronally advanced flap (CAF) with connective tissue graft(CTG) resulting from the de-epithelialization of a free gingival graft. In the test group (20 patients) a quadruple layer of PRF membrane will be placed over the palatal wounds; conversely, the control groups patients will be treated by an absorbable gelatin sponge. Patients will be monitored at 1, 2, 3 and 4 weeks after surgery for the complete re-epithelialization of the palatal wound (CWE), the alteration of sensibility (AS) around the wound area, the post-operative discomfort (D), and the changes of feeding habits (CFH) by a visual analogic scale (VAS) evaluation. Furthermore, the analgesics consumption and the existence of delayed bleeding from the palatal wound (DWB) during the first post-operative week will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* to have a single gingival recession to be treated by a mucogingival surgery intervention
* to be in good systemic health
* to have a good oral hygiene

Exclusion Criteria:

* no systemic diseases; no coagulation disorders; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation;
* no smoking habits;
* no periodontal surgery on the experimental sites;
* no inadequate endodontic treatment
* no tooth mobility at the site of surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Time needed to obtain a complete re epithelialization of the palatal wound | 4 weeks
  The primary outcome is to assess the time needed to obtain a complete re epithelialization of the palatal wound

CONTACTS AND LOCATIONS:
Overall Officials: michele paolantonio, Study Director — università G. D'annunzio Chieti-Pescara
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No